CLINICAL TRIAL: NCT05260788
Title: Feasibility of Spatially Registered Endoscopy for Mapping Bladder Mucosal Disease Into Radiation Planning Morphologic Imaging
Brief Title: Mapping 3D Bladder
Status: Withdrawn | Type: Observational
Why Stopped: Administrative issues.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-5338
Record Dates: First submitted 2022-01-28; First posted 2022-03-02 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cystoscopy — Standard of care cystoscopy procedure

SUMMARY:
This is a single centre, single arm feasibility study assessing the feasibility of using computer vision methods to recreate the 3D bladder shape and to then map the cystoscopy images onto this bladder shape. If feasible, this 3D reconstructed shape would be spatially registered to radiological images (CT, MR) that are then used during radiation treatment planning. This analysis would not be used for making any clinical treatment decisions on the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical suspicion or histologic diagnosis of bladder tumour suitable for endoscopic evaluation.
* Intention to treat using external beam radiation therapy as part of standard of care.
* Ability to provide written informed consent to participate in the study.

Exclusion Criteria:

* Prior complete or partial radiation therapy to bladder.
* Contraindications to radiation therapy as determined by the treating physician.
* Concurrent illness or condition that precludes subject from undergoing endoscopy or CT scanning.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion or histologic diagnosis of bladder tumour suitable for endoscopic evaluation and intent to treat using external beam radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Video recording of Cystoscopy | At study completion, up to 2 years
  To determine the feasibility of using bladder endoscopic video images to reconstruct the three-dimensional shape of the bladder based on computer visions methods that employ feature extraction and triangulation and to map the endoscopy images onto the recreated 3D surface.
Contouring of 3D bladder rendering | At study completion, up to 2 years
  To determine the feasibility of contouring the mucosal disease on the 3D bladder rendering.
Registering bladder shape | At study completion, up to 2 years
  To determine the feasibility of registering the bladder shape to a CT/MR scan of the patient using deformable shape methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada